CLINICAL TRIAL: NCT02506699
Title: Observational Study of the Analgesic Effect of Treatment With rTMS in Patients Suffering From Chronic Neuropathic Pain Refractory to Conventional Treatment and Monitored and Evaluated in Consultation Multidisciplinary Chronic Pain in Lower Normandy
Brief Title: Observational Study of the Analgesic Effect of Treatment With rTMS in Patients With Chronic Neuropathic Pain
Acronym: rTMSDOULNEURO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 13-025
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- analgesic effect of rTMS: Observe the analgesic effect of rTMS, reference method of noninvasive stimulation of the motor cortex validated by data from the literature and current practice, after 5 separate sessions a week apart, patients with neuropathic pain chronic, refractory to first and second-line treatments proposed in a multidisciplinary center specializing in chronic pain Lower Normandy.
  Interventions: Other: analgesic effect of rTMS

INTERVENTIONS:
Other: analgesic effect of rTMS

SUMMARY:
For ten years, rTMS, repetitive transcranial magnetic stimulation of the motor cortex, has found its place in the treatment of drug-resistant neuropathic pain. Patients relieved by some sessions may thereafter receive a chronic invasive stimulation via electrodes implanted through a neurosurgical procedure. This is common practice at the University Hospital of Caen and in different CHU with the proper equipment rTMS. It seems permissible to provide in our center only a non-invasive technique for patients challenged with brain surgery, since according to the various meta-analyzes the analgesic efficacy of rTMS seems to be correlated to the repetition of sessions.

Assessment centers and the treatment of pain allow a multidimensional assessment, bio-psycho-social of patients in order to optimize their management and experience efficiently analgesics first- and second-line.

We propose a study evaluating the analgesic efficacy of rTMS, in relevant stimulation parameters reproduced according to a literature review, during 3 months after 5 active sessions separated by one week apart, in 15 patients with neuropathic pain chronic refractory to treatment of first and second line, followed by multidisciplinary center specializing in chronic pain Lower Normandy. The quality of life will also be assessed by validated scales, and the results will be compared to the literature data.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 to 70 years with:

  1. Pain lasting for more than six months;
  2. Monitoring in CETD in Normandy;
  3. Having had a bio-psycho-social assessment and have been the subject of a multidisciplinary discussions recorded in the medical record;
  4. Presenting unilateral neuropathic pain, central or peripheral origin:

     * may affect the face,
     * upper limb,
     * or hémicorps but including at least the upper limb;
  5. With neuropathic pain screening test positive (≥ DN4 4/10);
  6. etiology objectified by further examinations (MRI, scanner, or EMG, PES MEP);
  7. Resistant to usual treatments: less than 50% improvement compared to the initial pain (EN or EVA) in patients who received an effective dose for treatment of first and a second intention.

Exclusion Criteria:

* Contraindications of rTMS:

  1. Brain implanted ferromagnetic material,
  2. Implanted neurostimulator (cortical and deep brain, spinal cord)
  3. Cochlear Implants
  4. Active epilepsy (seizures despite existence of a current treatment)
  5. Pacemakers
  6. Hearing loss or current taking ototoxic drugs (aminoglycosides, cisplatin)
* Pregnancy, breastfeeding, lack of effective contraception for patients of childbearing age
* Psychiatric illness decompensated
* Cancer pain and post-chemotherapy
* severe cognitive disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Neuropathic Pain
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
NPSI (Neuropathic Pain Symptom Inventory) | baseline and after 17 weeks
  Analysis of analgesic efficacy: evolution of NPSI (Neuropathic Pain Symptom Inventory), validated scale in monitoring neuropathic pain, and VAS (visual analogue scale), to fill once a week over a period of 17 weeks, from one week before the first session of rTMS until three months after the last rTMS session.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'évaluation et de traitement de la douleur (CETD), Caen, France